CLINICAL TRIAL: NCT06577870
Title: Immersive Sensory Projections: Evaluating the Impact of an Immersive Sensory Environment (Visual, Auditory and Olfactory) on Reducing the Overall Discomfort of Patients Hospitalized in the Resuscitation and Continuing Care Units
Brief Title: Immersive Sensory Projections for Hospitalized Patients
Acronym: IHP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Collaborators: Euraxi Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-A01322-45
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Hospitalism
MeSH Terms: interventions — Hospitalization; Critical Care

STUDY DESIGN:
Intervention Model Description: Multicenter, interventional, prospective, randomized, controlled study
Masking Description: Open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immersive sensory projections (Experimental): Patients will benefit from an immersive sensory environment in the hospital room. This IHP immersive sensory environment consists of the following elements:
  * light frescoes on the theme of nature, of the canopy type, diffused by a generative circadian cycle.
  * a soundtrack made up of nature sounds and sounds of life outside the hospital, broadcast in an immersive (moving sounds in the room), random (non-repetitive sounds over time) and generative way.
  * essential oils
  Interventions: Procedure: Hospitalization in intensive care or continuing care unit
- No immersive sensory projections (Active Comparator): Standard (control) group: Patients will not have any Immersion Health Project-type immersive sensory projection in the hospital room.
  Interventions: Procedure: Hospitalization in intensive care or continuing care unit

INTERVENTIONS:
Procedure: Hospitalization in intensive care or continuing care unit — Hospitalization in intensive care or continuing care unit for medical reasons or surgery, conscious or unconscious under mechanical ventilation. Resuscitation patients are then cared for in a continuing care unit.

SUMMARY:
The purpose of this study is to assess the impact of adding three sensory elements (visual, auditory, olfactory) on reducing discomfort in patients hospitalized in the intensive care unit/continuing care unit.

DETAILED DESCRIPTION:
The IHP trial is multicenter, interventional, prospective, randomized, controlled, open-label study.

The study population consists of adult patients hospitalized in an intensive care or continuing care unit for medical or surgical reasons, conscious or unconscious under mechanical ventilation.

All patients participating in the study will be managed according to usual practices in intensive care and continuing care units. All patients and their relatives will be monitored and supported by the medical team as in normal practice.

The study will be offered to the patient or a close relative/trusted person on admission to hospital.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years ;
* Patient hospitalized in intensive care or continuing care unit for an estimated minimum of 48 hours;
* Patient hospitalized for a medical indication (including in the pre-surgical phase) or in the post-surgical phase;
* Patient or support person who speaks and understands French, has understood the research procedures and is able to complete the questionnaires;
* For women of childbearing age (non-menopausal), even for those on contraception: negative pregnancy test (urinary); If positive: completed by a biological test;
* Patient or trusted support person having been informed and having signed an informed consent form to participate in the study.

Exclusion Criteria:

* Deaf or blind patient;
* Asthmatic patient with background treatment;
* Epileptic patient or known history of convulsion;
* Known allergy or intolerance to essential oils or to a component of essential oils;
* Patient transferred from another intensive care unit;
* Protected patient (under legal protection, or deprived of liberty by judicial or administrative decision);
* Breast-feeding or pregnant women;
* Patient or support person unable to understand information relating to the study (linguistic, psychological, cognitive, etc.);
* Unconscious patient with no relative or support person present;
* Homeless patient;
* Patient with known severe psychiatric illness such as chronic hallucinatory psychosis or paranoid syndrome;
* Patient participating in or being excluded from another clinical trial;
* Patient not covered by a social security scheme.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
REAnimation Patient Discomfort Questionnaire | 2 months
  Overall score on the REAnimation Patient Discomfort Questionnaire at the end-of-study visit

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé Jacques Cartier, Massy, France

IPD SHARING:
Plan to Share IPD: No